CLINICAL TRIAL: NCT04660617
Title: A Multi-omics Study of Metastatic Prostate Cancer (MOSMPCA)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Hao Zeng, Vice director of the department of urology, West China Hospital
Other Study IDs: MOSMPCA
Record Dates: First submitted 2020-11-01; First posted 2020-12-09 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Prostate Cancer Metastatic
Keywords: Genomic sequencing; Transcriptome sequencing; Epigenetics; Metabonomics; Immunohistochemical; Multi-omics Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators plan to perform multi-omics technologies, including genomic, transcriptomic, epigenomic and proteomic methods, in patients with metastatic prostate cancer, aiming at uncovering the mechanism of the tumor progression, identifying distinct tumor subtypes and finding new treatment targets.

DETAILED DESCRIPTION:
Prostate cancer is the commonest malignancy and the second leading cause of tumor-related death among males worldwide. Though patients with early stage prostate cancer can obtain satisfactory therapeutic efficacy from radical prostatectomy or radiotherapy, the prognosis of men with metastatic prostate cancer (mPCa), especially metastatic castration-resistant prostate cancer (mCRPC), is still poor. Recent years have witnessed the rapid development of the high-throughput technologies, including genomic, transcriptomic, epigenomic and proteomic methods. These techniques are promising in uncovering the mechanism of the tumor progression, identifying distinct tumor subtypes and finding new treatment targets.

In the current prospective study, the investigators plan to perform multi-omics technologies in patients with mPCa, aiming at uncovering the mechanism of the tumor progression, identifying distinct tumor subtypes and finding new treatment targets.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmation of prostate cancer
* Age: ≥40 years old
* Bone or visceral metastatic disease confirmed by image examination.
* Written informed consent

Exclusion Criteria:

* Patients harbouring other types of cancer besides prostate cancer

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male patient can enter this study
Study Population: Patients with primary metastatic prostate cancer are potentially eligible for the current study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Genetic profiling results | From baseline (initial diagnosis of PCa), until study completion (48 months)
  Mutation identified via whole-genome sequencing will be recored.
Transcriptional profiling results | From baseline (initial diagnosis of PCa), until study completion (48 months)
  Determining the transcriptomic information of metastatic prostate cancer by performing whole transcriptome sequencing
Epigenomic profiling results | From baseline (initial diagnosis of PCa), until study completion (48 months)
  Determining the epigenomic status of specific genes by performing DNA-methylation sequencing

SECONDARY OUTCOMES:
Protein expression results | From baseline (initial diagnosis of PCa), until study completion (48 months)
  Determing the expression status of centain proteins by performing immunohistochemistry in prostate biopsy specimen

CONTACTS AND LOCATIONS:
Overall Officials: Hao Zeng, Dr., Principal Investigator — West China Hospital

IPD SHARING:
Plan to Share IPD: Undecided